CLINICAL TRIAL: NCT02464085
Title: Characterising Arm Recovery in People With Severe Stroke
Acronym: CARPSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H15-00083
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Neuroplastic change; Longitudinal; Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Longitudinal evaluation of recovery: Stroke survivors with subacute and severe upper limb disability
  Interventions: Other: Longitudinal evaluation of recovery

INTERVENTIONS:
Other: Longitudinal evaluation of recovery — Stroke survivors will be assessed at four time frames post stroke to evaluate neuroplastic and clinical changes in arm recovery over the first 12-months post stroke.

SUMMARY:
The main goal of this program of research is to advance our understanding of how the severely damaged brain changes over the first 12-months post stroke. The investigators will determine 'who recovers', 'who does not recover', and 'why'

DETAILED DESCRIPTION:
The main goal of this program of research is to advance our understanding of how the severely damaged brain changes over the first 12-months post stroke. The prevalence and severity of stroke related arm disability is increasing and the prospect of optimal recovery is poor. Studies have demonstrated that stroke survivors with severe disability lack early indicators (<7-days to <1-month post-stroke) of a good prognosis, such as active movement at the shoulder and wrist and integrity of the corticospinal tract. This has propagated the clinical belief that this cohort are unlikely to functionally benefit from rehabilitation efforts. However, it is possible that indicators of potential for recovery - either neuroanatomical or clinical - may present in individuals with severe stroke later, that is beyond the early time-period. Indeed, there is increasing evidence of the potential for ongoing improvements in motor performance in response to intensive interventions that are undertaken 6-months or more post-stroke. This therefore, implies that there is some degree of untapped recovery potential. However, as very few studies have longitudinally explored the potential indicators of recovery in a severe cohort, the dynamic capacity of the severely damaged remains unknown. Thus, there is a need to determine 'who recovers', 'who does not recover', and 'why' to be able to promote optimal arm recovery in people with severe impairment after stroke. We will assess stroke survivors <4-weeks, 3-months, 6-months and 12-months post stroke using a range of neuroimaging and clinical outcome measures. The findings from this study will build the foundations for more personalized health care options for people with severe arm impairment post stroke.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 90 years;
* sustained their first stroke;
* demonstrate subacute (<1 month) and severe upper limb motor deficits (defined by a SAFE [shoulder abduction and finger extension] score of <5 out of 10 points); and
* can follow single stage commands

Exclusion Criteria:

* neurological condition other than stroke e.g., Parkinson's disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors with subacute and severe upper limb disability will be evaluated longitudinally.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
3T Magnetic Resonance Imaging (MRI) | up to 12-months
  Determine the structural and functional connectivity of the brain using diffusion weighted imaging, resting state-functional magnetic resonance imaging and myelin water fraction imaging.

SECONDARY OUTCOMES:
Shoulder abduction and finger extension (SAFE) | 12-months
  Measurement of upper limb strength
Fugl-Meyer Assessment (arm and sensory) | <4wks, 3-months, 6-months, 12-months
  Measurement of upper limb impairment
Motor Assessment Scale items 6,7,8 | <4wks, 3-months, 6-months, 12-months
  Measurement of upper limb activity
REACH (Rating of Everyday Arm Use in the Community and Home) | <4wks, 3-months, 6-months, 12-months
  Self-report measure of everyday arm use
Accelerometry | <4wks, 3-months, 6-months, 12-months
  Measurement of real world arm use (activity count) over a 7-day period at each time frame
PASS (Postural Assessment Scale for Stroke patients) | <4wks, 3-months, 6-months, 12-months
  Measurement of balance (static and dynamic) and lower limb functional tasks
10-metre walk test | <4wks, 3-months, 6-months, 12-months
  Measurement of walking ability
Montreal Cognitive Assessment (MoCA) | <4wks, 3-months, 6-months, 12-months
  Measurement of cognitive impairment after stroke
Dose of upper limb training | <4wks, 3-months, 6-months, 12-months
  Dose in minutes of passive, active, functional or sensory upper limb tasks performed over a 7-day period at each time frame
National Institute of Stroke Severity Scale | <4-weeks
  Characterise stroke severity
Oxfordshire Bamford Classification | <4-weeks
  Characterise stroke type
Myelin water fraction imaging (WMI) | <4wks, 3-months, 6-months, 12-months
  Determine the myelin content within the brain
Meaningful arm recovery questionnaire | <4wks, 3-months, 6-months, 12-months
  Explore the stroke survivor's perception of meaningful recovery of their upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Boyd, PT PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hayward KS, Lohse KR, Bernhardt J, Lang CE, Boyd LA. Characterising Arm Recovery in People with Severe Stroke (CARPSS): protocol for a 12-month observational study of clinical, neuroimaging and neurophysiological biomarkers. BMJ Open. 2018 Nov 25;8(11):e026435. doi: 10.1136/bmjopen-2018-026435. PMID 30478130